CLINICAL TRIAL: NCT00606788
Title: Comparison of Computer-Driven Protocolized Weaning With Physician-Directed Weaning in Surgical Intensive Care Unit (ICU) Patients
Brief Title: Therapy Study of Automated Protocolized vs. Physician-Directed Non-Protocolized Weaning
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated that sample size of study patients had to be highly increased to obtain significant outcomes.
Sponsor: University of Luebeck (Other)
Responsible Party: Prof. Dr. med. Elke Muhl, Department of Surgery and Surgical Intensive Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Luebeck 0001
Record Dates: First submitted 2008-01-16; First posted 2008-02-05 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Neoplasms; Musculoskeletal Diseases; Digestive System Diseases; Respiratory Tract Diseases; Cardiovascular Diseases
Keywords: randomized clinical trials; intensive care; mechanical ventilation; ventilator weaning; clinical protocols; therapy, computer-assisted; humans; various surgical diseases requiring mechanical ventilation over 24 hours
MeSH Terms: conditions — Neoplasms; Musculoskeletal Diseases; Digestive System Diseases; Respiratory Tract Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AW (Active Comparator): Patients received computer-driven protocolized weaning (= Automated Weaning)
  Interventions: Device: SmartCare/PS (Automated Weaning)
- CW (Active Comparator): Patients received physician-directed non-protocolized weaning (= Conventional Weaning)
  Interventions: Procedure: Conventional weaning

INTERVENTIONS:
Device: SmartCare/PS (Automated Weaning) — Patients received computer-driven protocolized weaning
  Other Names: SmartCare/PS (Draeger Medical AG & Co. KG, Luebeck, Germany)
  Arms: AW
Procedure: Conventional weaning — Patients received physician-directed non-protocolized weaning
  Arms: CW

SUMMARY:
The purpose of this study was to determine whether computer-driven protocolized weaning is superior to physician-directed non-protocolized weaning in over-24-hours-ventilated surgical intensive care unit (ICU) patients. The main hypothesis was that weaning duration differs between both methods. Secondary hypotheses were that reintubation rate, duration of mechanical ventilation, intensive care unit (ICU) length of stay and workload for physicians and nurses differ between both methods.

DETAILED DESCRIPTION:
Since long-term mechanical ventilation is affiliated with a bunch of complications, weaning affected patients from ventilation as soon as possible is a crucial point. In this context automated computerized systems have become a torchbearer. These systems are expected to expedite the weaning process, reduce the duration of mechanical ventilation and ICU length of stay of a given patient in comparison to conventional physician-directed weaning. A multicenter randomized trial by Lellouche et al supported these theories, using a computer-driven system to regulate Pressure Support Ventilation (PSV). This system is now commercially available as SmartCare/PS (Draeger Medical AG & Co. KG, Luebeck, Germany).

The purpose of the study on hand was to find out whether the results reported before could be repeated in a broad, surgical ICU patient group. Study design was chosen similar. In addition we investigated the workload for physicians and nurses in both study arms which has not been conducted before.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation > 24 hours
* intubation OR tracheostomy
* informed consent
* 35 - 200 kg bodyweight (77,2 - 440,9 lb)
* Ramsay-Score < 3
* spontaneous breathing at a PEEP of < 10 cm H2O
* sufficient arterial oxygenation (paO2 > 55 mmHg or SaO2 > 90%)
* haemodynamic stability (< 5 µg/kg/min Dopamine)
* body temperature (rectal) max. 39 °C / 102.2 °F
* hemoglobin > 7 g/dl
* pH > 7,2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Estimated); Study Completion 2007-02 (Estimated)

PRIMARY OUTCOMES:
weaning duration | measured in days

SECONDARY OUTCOMES:
reintubation rate | expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Elke Muhl, Prof. Dr. med., Principal Investigator — University of Luebeck
Locations (1):
- UKSH Campus Luebeck, Department of Surgery and Surgical Intensive Care, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Lellouche F, Mancebo J, Jolliet P, Roeseler J, Schortgen F, Dojat M, Cabello B, Bouadma L, Rodriguez P, Maggiore S, Reynaert M, Mersmann S, Brochard L. A multicenter randomized trial of computer-driven protocolized weaning from mechanical ventilation. Am J Respir Crit Care Med. 2006 Oct 15;174(8):894-900. doi: 10.1164/rccm.200511-1780OC. Epub 2006 Jul 13. PMID 16840741